CLINICAL TRIAL: NCT05102162
Title: Beta-lactam Continuous Versus Intermittent Infusion and Associated Bacterial Resistance and Therapy Outcomes in Critically Ill Patients With Severe Pneumonia
Brief Title: BL Infusion Trial:Beta-lactam Continuous Versus Intermittent Infusion and Associated Bacterial Resistance and Therapy Outcomes in Critically Ill Patients With Severe Pneumonia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment.
Sponsor: University of Florida (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202101979 -A; OCR41108 (Other: UF OnCore)
Record Dates: First submitted 2021-10-29; First posted 2021-11-01 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-05

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Cefepime; Meropenem; Piperacillin; Tazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Continuous Antibiotic Dose Over 24 hours Arm (Active Comparator): Subjects will be receiving a continuous dose of antibiotic prescribed by their doctor for the duration they choose.
  Interventions: Drug: Cefepime, Meropenem, or Piperacillin/Tazobactam
- Intermittent Antibiotic Dose Over 30 minutes (Active Comparator): Subjects will be receiving an intermittent dose of antibiotic prescribed by their doctor for the duration they choose.
  Interventions: Drug: Cefepime, Meropenem, or Piperacillin/Tazobactam

INTERVENTIONS:
Drug: Cefepime, Meropenem, or Piperacillin/Tazobactam — A 1:1 randomization scheme based on the infusion duration (continuous over 24 hours or intermittent over 30 minutes) with stratification based on the beta-lactam prescribed (cefepime, meropenem, or piperacillin/tazobactam)
  Other Names: Maxipime, Merrem
  Arms: Continuous Antibiotic Dose Over 24 hours Arm
Drug: Cefepime, Meropenem, or Piperacillin/Tazobactam — A 1:1 randomization scheme based on the infusion duration (continuous over 24 hours or intermittent over 30 minutes) with stratification based on the beta-lactam prescribed (cefepime, meropenem, or piperacillin/tazobactam)
  Other Names: Maxipime, Merrem
  Arms: Intermittent Antibiotic Dose Over 30 minutes

SUMMARY:
The study plans to randomize a total of 240 patients infected with Gram-negative bacterial pneumonia to receive beta-lactam (meropenem, cefepime, or piperacillin/tazobactam) continuous or intermittent infusion and collect baseline and regular follow-up respiratory cultures to assess the development of new resistance. The investigators will measure beta-lactam concentration to assess the impact of drug exposure on the bacterial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ICU with severe pneumonia (IDSA/ATS 2016/2019): presence of signs, symptoms and confirmatory chest imaging consistent with pneumonia (e.g. fever, cough and pulmonary infiltrate by chest radiograph)
* Age ≥18 years
* Positive respiratory culture (with or without an initial positive rapid identification test and/or Gram stain) for Gram-negative bacteria including, but not limited to, P. aeruginosa, K. pneumoniae, E. coli, S. marcescens, H. influenzae, Enterobacter spp., M. catarrhalis, A. baumannii, Achromobacter spp., P. mirabilis, and/or B. cepacia
* Received within the last 72 hours or will receive meropenem, cefepime, or piperacillin/tazobactam therapy

Exclusion Criteria:

* Pregnancy
* Prisoners
* Allergy to the beta-lactams to be administered in this study
* On renal replacement therapy at the time of randomization
* Baseline culture resistant to the beta-lactams in the study
* COVID patients enrolled in other trials

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Peloquin, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
Started | 19 | 16
Completed | 5 | 13
Not Completed | 14 | 3
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Baseline cultures negative | 4 | 2
Not completed — <72 Hours on study beta-lactam | 7 | 0
Not completed — Baseline cultures resistant to all study beta-lactams | 0 | 1

BASELINE CHARACTERISTICS:
Population: Each participant that was unenrolled from the study was assessed to determine if the data could be used in the final analysis. 17 participants completed the study and we unenrolled 18 participants. However, we were able to use the data from 1 participant in the final analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes | Total
Number analyzed (Participants) | 5 | 13 | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [49 to 74] | 69 [61 to 73] | 69 [58 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 4 | 8 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 3 | 9 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 13 | 18
Weight (kg) [Median (Inter-Quartile Range); unit: kg] | 103.4 [63.7 to 120] | 61.6 [51.4 to 89.1] | 75.3 [55.1 to 100.7]
Serum Creatinine (mg/dL) [Median (Inter-Quartile Range); unit: mg/dL] | 1.21 [0.66 to 2.16] | 0.67 [0.54 to 1.09] | 0.76 [0.59 to 1.23]
Creatinine clearance (mL/min) [Median (Inter-Quartile Range); unit: mL/min] | 92 [77.7 to 222.8] | 83.7 [69.4 to 105.4] | 86.7 [69.7 to 114.9]
BMI (kg/m^2) [Median (Inter-Quartile Range); unit: kg/m^2] | 31.6 [26.4 to 42.9] | 22.4 [19.2 to 30.7] | 24.8 [20.7 to 32.6]
Height (m) [Median (Inter-Quartile Range); unit: meters] | 1.75 [1.70 to 1.8] | 1.65 [1.65 to 1.73] | 1.68 [1.65 to 1.76]
Beta-Lactam at Randomization [Count of Participants; unit: Participants]
  Cefepime | 4 | 7 | 11
  Meropenem | 0 | 2 | 2
  Piperacillin/tazobactam | 1 | 4 | 5

OUTCOME MEASURES:

1. Primary Outcome: Gram-negative Bacterial Resistance Emergence Between Patients Treated With Continuous and Intermittent Infusion Beta-lactam Regimens
Description: Bacterial resistance is defined as new numeric increases (>/=2 fold) in the bacterial MIC during the follow-up period compared to the baseline when starting beta-lactam therapy. MICs were collected from respiratory samples and compared from study enrollment to end of the follow-up period for at least a 2 fold increase in MIC.
Time Frame: 4 weeks
Population: The number of participants included in the analysis was 18. However, for the primary outcome measure, the bacteria isolates were analyzed for emergence of resistance. We were able to include 18 isolates in the intermittent infusion arm and 8 in the continuous infusion arm.
Measure: Number; unit: Bacteria isolates
Units Other Than Participants: Bacteria isolates
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
Number analyzed (Participants) | 5 | 13
Number analyzed (Bacteria isolates) | 8 | 18
Bacteria isolates | 4 | 8

2. Secondary Outcome: Superinfection Between Patients Treated With Continuous and Intermittent Infusion Beta-lactam Regimens.
Description: Superinfection is defined as the growth of resistant Gram-negative bacteria during the follow-up period which was not isolated in baseline culture. Respiratory cultures during the follow up period were assessed for Gram-negative isolates resistant to the beta-lactams of interest that were not present in the initial respiratory cultures.
Time Frame: 4 weeks
Population: The number of participants included in the analysis was 18. However, for superinfection, the bacteria isolates were analyzed. We were able to include 18 Gram-negative isolates in the intermittent infusion arm and 8 Gram-negative isolates in the continuous infusion arm.
Measure: Number; unit: Bacteria isolates
Units Other Than Participants: Bacteria Isolates
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
Number analyzed (Participants) | 5 | 13
Number analyzed (Bacteria Isolates) | 8 | 18
Bacteria isolates | 0 | 0

3. Secondary Outcome: Microbiologic Eradication Between Patients Treated With Continuous and Intermittent Infusion Beta-lactam Regimens
Description: Microbiologic eradication is defined as the absence of bacterial growth during the follow-up period with no subsequent positive culture from any site. Respiratory cultures during the follow up period were assessed for the absence of bacterial growth.
Time Frame: 4 weeks
Population: For microbiologic eradication, the bacteria isolates were analyzed. We were able to include 18 Gram-negative isolates in the intermittent infusion arm and 8 Gram-negative isolates in the continuous infusion arm.
Measure: Number; unit: Bacteria isolates
Units Other Than Participants: Bacteria Isolates
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
Number analyzed (Participants) | 5 | 13
Number analyzed (Bacteria Isolates) | 8 | 18
Bacteria isolates | 1 | 4

4. Secondary Outcome: Clinical Cure at Day 7 of Therapy Between Patients Treated With Continuous and Intermittent Infusion Beta-lactam Regimens
Description: Clinical cure is the resolution of infection-related symptoms at day 7 of therapy, including normalization of body temperature and white blood cell (WBC) count and taking the patient off mechanical ventilation or vasopressors, and non-initiation of a new antibiotic within 48 hours of stopping the original antibiotic.
Time Frame: 7 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
Number analyzed (Participants) | 5 | 13
Participants | 0 | 5

5. Secondary Outcome: Clinical Cure at the End of Therapy Between Patients Treated With Continuous and Intermittent Infusion Beta-lactam Regimens
Description: Clinical cure is the resolution of infection-related symptoms at the end of therapy, including normalization of body temperature and white blood cell (WBC) count and taking the patient off mechanical ventilation or vasopressors, and non-initiation of a new antibiotic within 48 hours of stopping the original antibiotic. End of therapy could occur up to 4 weeks after enrollment.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
Number analyzed (Participants) | 5 | 13
Participants | 3 | 8

6. Secondary Outcome: Mortality Between Patients Treated With Continuous and Intermittent Infusion Beta-lactam Regimens
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
Number analyzed (Participants) | 5 | 13
Participants | 2 | 2

7. Secondary Outcome: Hospital Length of Stay Between Patients Treated With Continuous and Intermittent Infusion Beta-lactam Regimens.
Time Frame: 4 weeks (may extend beyond depending on patient length of stay in hospital)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
Number analyzed (Participants) | 5 | 13
Days | 27 [12 to 32] | 18 [13 to 32]

8. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay Between Patients Treated With Continuous and Intermittent Infusion Beta-lactam Regimens
Time Frame: 4 weeks (may extend beyond depending on patient length of stay in ICU)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
Number analyzed (Participants) | 5 | 13
Days | 23 [7 to 26] | 9 [6 to 17]

9. Secondary Outcome: Percent of Time Free Drug Concentrations Remain Above the Minimum Inhibitory Concentration (%fT>MIC) in the Dosing Interval Between Patients Treated With Continuous and Intermittent Infusion Beta-lactam Regimens
Description: Beta-lactam bactericidal efficacy depends upon the percentage of time that free drug concentrations remain above the minimum inhibitory concentration (%fT>MIC) of the pathogen within the dosing interval. Pre-clinical animal studies demonstrate 40-70% fT>MIC is needed for adequate bacterial killing. However, clinical studies suggest higher exposures may be needed, potentially 100%fT>MIC to 100%fT>4xMIC. Patients had beta-lactam concentrations measured as part of therapeutic drug monitoring. Drug exposures were determined using a Bayesian-based software. Infusion arms were compared to determine if %fT>MIC was different between infusion arms.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage of time
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
Number analyzed (Participants) | 5 | 13
Percentage of time | 100 [100 to 100] | 100 [94 to 100]

10. Secondary Outcome: Percent of Time Free Drug Concentrations Remain Above Four Multiples of the Minimum Inhibitory Concentration (%fT>4xMIC) in the Dosing Interval Between Patients Treated With Continuous and Intermittent Infusion Beta-lactam Regimens
Description: Beta-lactam bactericidal efficacy depends upon the percentage of time that free drug concentrations remain above the minimum inhibitory concentration (%fT>MIC) of the pathogen within the dosing interval. Pre-clinical animal studies demonstrate 40-70% fT>MIC is needed for adequate bacterial killing. However, clinical studies suggest higher exposures may be needed, potentially 100%fT>MIC to 100%fT>4xMIC. Patients had beta-lactam concentrations measured as part of therapeutic drug monitoring. Drug exposures were determined using a Bayesian-based software. Infusion arms were compared to determine if %fT>4xMIC was different between infusion arms.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: Percentage of time
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
Number analyzed (Participants) | 5 | 13
Percentage of time | 100 [50 to 100] | 100 [58 to 100]

ADVERSE EVENTS:
Time Frame: Each participant was monitored for adverse events for the duration of enrollment in the study (up to 4 weeks).
Arm/Group | Continuous Antibiotic Dose Over 24 Hours Arm | Intermittent Antibiotic Dose Over 30 Minutes
All-Cause Mortality (participants affected / at risk) | 2/19 | 2/16
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/16
Other Adverse Events (participants affected / at risk) | 0/19 | 0/16

LIMITATIONS AND CAVEATS:
* Early termination leading to a small sample size and under-powered study.
* Repeat positive cultures may have been due to colonization and not active infection, especially in participants demonstrating clinical cure prior to repeat cultures.
* This study used MICs, which are generally accepted to have variability with repeat assessments, potentially up to 200% or more.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT05102162/Prot_SAP_000.pdf
  • Informed Consent Form (2022-11-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT05102162/ICF_001.pdf